CLINICAL TRIAL: NCT04618393
Title: A Phase I/II Trial of EMB-02, a Bi-specific Antibody Against PD-1 and LAG-3, in Patients With Advanced Solid Tumors
Brief Title: A Study of EMB-02 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company's resource optimization and product's development change
Sponsor: Shanghai EpimAb Biotherapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB02X101
Record Dates: First submitted 2020-10-18; First posted 2020-11-05 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors
Keywords: Phase I/II; Bispecific antibody; PD-1; LAG-3; EMB-02; Immuno-oncology; dose escalation; cohort expansion; Neoplasms; Neoplasm Metastasis; advanced solid tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Dose escalation followed by Cohort Expansion Phase at the RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EMB-02 (Experimental): In Phase I part: participants enrolled in the different time will receive EMB-02 once weekly (IV) at different ascending dose levels.
  In Phase II part: participants will receive EMB-02 once weekly (IV) at previously defined RP2D.
  Interventions: Biological: EMB-02

INTERVENTIONS:
Biological: EMB-02 — EMB-02 is a FIT-Ig® bispecific antibody against PD-1 and LAG-3.

SUMMARY:
The primary purpose of this study is to identify the recommended Phase 2 dose(s) (RP2Ds) and schedule assessed to be safe for EMB-02 and to characterize the safety and tolerability of EMB-02 at the RP2Ds. Pharmacokinetics (PK), immunogenicity, and the anti-tumor activity of EMB-02 will also be assessed.

DETAILED DESCRIPTION:
This is a Phase I/II, multi-center, open label, multiple-dose, first in human study, designed to assess safety and tolerability, and to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dos(s)e (RP2D[s]) for EMB-02 in patients with advanced solid tumors. Pharmacokinetics, pharmacodynamics, immunogenicity, and response will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Phase I: Patients with histologically or cytologically confirmed locally advanced/metastatic solid tumors and have failed (progressed on, or are intolerant of) standard therapies. Moreover, the disease should be measurable or evaluable per RECIST v1.1
* Phase II Cohort A: Patients with histologically or cytologically confirmed locally advanced/metastatic melanoma, excluding uveal melanoma. > 1 prior therapy, including prior treatment with PD-1/L1(mandatory) and/or CTLA-4 inhibitors(optional). And the disease is measurable or evaluable per RECIST v1.1
* Archival tumor samples available for retrospective analysis or biopsy will be taken.
* ECOG performance status 0 or 1 for phase I, and ≤2 for phase II; life expectancy > 3 Months
* Adequate organ function to participate in the trial.
* Recovery from adverse events (AEs) related to prior anticancer therapy.
* Highly effective contraception

Exclusion Criteria:

* Patients who have active autoimmune disease or history of autoimmune disease
* History of severe irAE.
* History of severe allergic reactions
* Use of systemic corticosteroids.
* Symptomatic central nervous system metastases.
* Patients with cardiac dysfunction
* Uncontrolled diabetes mellitus with hemoglobin A1c > 8% (via medical history)
* Prior treatment with a LAG-3 inhibitor
* Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study treatment;
* Prior organ or stem cell/bone marrow transplant.
* Concurrent malignancy < 5 years prior to entry.
* Patients with active infections.
* Major surgery < 4 weeks or minor surgery < 2 weeks prior to study treatment
* Live virus vaccines < 30 days prior to screening
* Pregnant or breast-feeding females
* Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment
* Any other serious underlying medical conditions
* Abuse on alcohol, cannabis- derived products or other drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events as assessed by CTCAE V5.0 | Screening up to follow-up (30 days after the last dose)
  Incidence and severity of AE.
Incidence of serious adverse events (SAE) | Screening up to follow-up (30 days after the last dose)
  Incidence of SAE.
Incidence of dose interruptions | Screening up to follow-up (30 days after the last dose)
  Incidence of dose interruptions of EMB-02 during treatment as a measure of tolerability.
Dose intensity | Screening up to follow-up (30 days after the last dose)
  Actual amount of drug taken by patients divided by the planned amount.
The incidence of DLTs during the first cycle of treatment. | First infusion to the end of Cycle 1 (each cycle is 28 days)
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and are specifically defined in study protocol.
Antitumor activity(Objective Response Rate (ORR) | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Measured by RECIST 1.1, only applicable in Phase II part

SECONDARY OUTCOMES:
Area under the serum concentration-time curve (AUC) of EMB-02 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (AUC).
Maximum serum concentration (Cmax) of EMB-02 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Cmax)
Trough concentration (Ctrough) of EMB-02 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Ctrough)
Average concentration over a dosing interval (Css, avg)of EMB-02. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Css, avg).
Terminal half-life (T1/2) of EMB-02 | Through treatment until EOT visit, expected average 6 months.
  Blood samples for serum PK analysis will be obtained (T1/2)
Systemic clearance (CL) of EMB-02 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (CL).
Steady state volume of distribution (Vss) of EMB-02 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Vss).
Progression free survival (PFS) of EMB-02 as assessed by RECIST 1.1 | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Preliminary anti-tumor activity of EMB-02 will be obtained (PFS).
Duration of response of EMB-02 as assessed by RECIST 1.1 | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Preliminary anti-tumor activity of EMB-02 will be obtained (DOR).
Incidence and titer of anti-drug antibodies stimulated by EMB-02 | Up to End of Treatment Follow Up Period (30 days after the last dose)
  Antibodies to EMB-02 will be assessed to evaluate potential immunogenicity.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - University of Colorado Health Medical Group, Colorado Springs, Colorado
  - Prisma Health-Upstate, Greenville, South Carolina
- Australia (3):
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Monash Health, Clayton, Victoria
  - Peninsula & South Eastern Haematology & Oncology Group (PASO), Frankston, Victoria
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The first Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - HanDan Central Hospital, Handan, Hebei
  - HeNan Provincial People's Hospital, Zhengzhou, Henan
  - SuiNing Central Hospital, Suining, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Day D, Ganju V, Chung K, Si L, Mao L, Aghmesheh M, Hoyer R, Brewin K, Zeng S, Zhang M, Lu Q, Jiang C, Ren F, Zhu Y, Guo J. First-in-human phase I study of EMB-02, a bispecific antibody targeting PD-1 and LAG-3 in patients with advanced solid tumors. Br J Cancer. 2025 Jun;132(10):905-912. doi: 10.1038/s41416-025-02990-x. Epub 2025 Apr 15. PMID 40234667
- [Derived] Jiang C, Ren F, Zhang M, Lu Q, Zeng S, Yang G, Zhu Y. Using Pharmacokinetic and Pharmacodynamic Analysis to Optimize the Dosing Regimens of Fanastomig (EMB-02) in Patients With Advanced Solid Tumors. CPT Pharmacometrics Syst Pharmacol. 2025 May;14(5):975-986. doi: 10.1002/psp4.70011. Epub 2025 Mar 11. PMID 40067130